CLINICAL TRIAL: NCT01452438
Title: Post-licensure Observational Safety Surveillance Study of Quadrivalent Meningococcal ACWY Conjugate Vaccine MenACWY-CRM (Menveo) Vaccination in Children 2 Through 10 Years of Age
Brief Title: Safety Surveillance of MenACWY-CRM Vaccine in Children
Status: Completed | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V59_54OB
Record Dates: First submitted 2011-09-29; First posted 2011-10-14 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Meningococcal Disease
Keywords: observational; serogroup A, B, Y, W; meningococcal meningitis; meningococcal vaccines; safety; MenACYW-CRM; post-marketing; children
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal | interventions — MenACWY-CRM vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- MenACYW-CRM vaccinated children: All children between the age of 2 to 10 years old who have received of MenACYW-CRM vaccine during the study period.
  Interventions: Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenACWY-CRM — MenACYW-CRM vaccination received as part of routine clinical care and as registered in the vaccine records.

SUMMARY:
The purpose of this study is to summarize the occurrence of incident serious medically attended events and events of interest up to 1 year following MenACWY-CRM vaccination administered as part of routine clinical care. This US FDA post-marketing commitment study is an open-label, descriptive, epidemiological safety surveillance study of MenACWY-CRM vaccine in subjects 2 to 10 years of age within a large US Healthcare Maintenance Organization. The 26 events of interest are events commonly evaluated in vaccine safety studies and include certain neurological, immunological, vascular, musculoskeletal and hematologic disorders. All events are collected retrospectively.

DETAILED DESCRIPTION:
This is an observational study, vaccines administration and data that is collected is only as part of routine clinical care. Vaccinated subjects are not actively recruited.

Events of Interest: Diabetes Mellitus, Rheumatoid arthritis, Idiopathic Thrombocytopenic Purpura, Iridocyclitis, Acute glomerulonephritis, Nephrotic syndrome, Grave's disease, Autoimmune hemolytic anemia, Myasthenia Gravis, New onset asthma, Allergic urticaria, Anaphylaxis, Meningococcal Disease, Intentional Injury

ELIGIBILITY:
Inclusion Criteria:

* Registered with the HMO for at least 6 months prior to vaccination.
* Between the ages of 2 and 10 years (inclusive - i.e. has not reached their 11th birthday) at the time of the vaccination.
* Received any MenACWY-CRM vaccination during the vaccination period at the participating centers.

Exclusion Criteria:

* None

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population is selected from the Health Maintenance Organization population of the Kaiser Permanente Southern California (KPSC) HMO in Pasadena, CA, USA.
Sampling Method: Non-Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Timing relative to vaccination date (mean days (SD)) for all serious medically attended events and events of interest | Observational period of 1 year following date of vaccination of that individual.
Frequency (n, %) for all serious medically attended events and events of interest | Observational period of 1 year following date of vaccination of that individual.
Incidence (n per person years, 95% CI) for all serious medically attended events and events of interest | Observational period of 1 year following date of vaccination of that individual.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Kaiser Permanente South California, Pasadena, California, United States

REFERENCES:
- [Derived] Tartof SY, Sy LS, Ackerson BK, Hechter RC, Haag M, Slezak JM, Luo Y, Fischetti CA, Takhar HS, Miao Y, Solano Z, Jacobsen SJ, Tseng HF. Safety of Quadrivalent Meningococcal Conjugate Vaccine in Children 2-10 Years. Pediatr Infect Dis J. 2017 Nov;36(11):1087-1092. doi: 10.1097/INF.0000000000001696. PMID 28719502